CLINICAL TRIAL: NCT03984669
Title: (1,3)-Béta-D-Glucan Levels at Diagnosis of Juvenile Idiopathic Arthritis and Its Correlation With Activity's Disease : a Cohort Sudy
Acronym: BDG -JIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2018_843_0036
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: juvenile idiopathic arthritis; (1,3)-beta-D-glucan; children; inflammatory status; intestinal microbiota; activity od the disease
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Biological Assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: The Juvenile Disease Activity Score (JADAS) — The JADAS includes the following four measures: physician's global assessment of disease activity, measured on a 0-10 visual analog scale (VAS) where 0 = no activity and 10 = maximum activity; parent global assessment of well-being, measured on a 0-10 VAS where 0 = very well and 10 = very poor; the erythrocyte sedimentation rate (ESR), normalized to a 0 to 10 scale; and a count of joints with active disease.
Biological: (1-3)-ß-D-Glucan (BDG) assay (Fungitell) — Evaluation of the (1,3)-Beta-D-Glucans level in patients with JIA and correlation of the higher serum BDG levels with JIA activity of disease, comparatively with usual markers

SUMMARY:
Juvenile idiopathic arthritis (JIA) is the most common pediatric rheumatic disease of childhood. Most children still experience prolonged periods of active disease, however, there is still lack of effective and specific markers for early diagnosis of relapse. The pathogenesis of JIA is thought to be the result of a combination of host genetic and environmental triggers and The microbiota is a potential contributing factor to the development of the disease. (1-3)-ß-D-Glucan (BDG), a component of most fungal cell walls, possess immunomodulatory activities. Latest studies demonstrate that it acts as a trigger for autoimmune arthritis in adult. However the relation with JIA is not clearly defined. The objective of this study was to evaluate the (1,3)-Béta-D-Glucans level in patients with JIA and whether higher serum BDG levels are correlated with JIA activity of disease, comparatively with usual markers.

ELIGIBILITY:
Inclusion Criteria:

* All patients under the age of 18 years with JIA's disease
* followed at the CHU Amiens (French University hospital)
* signed parent consent form

Exclusion Criteria:

* lack of consent from parents or patient

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Measure of (1,3)-Beta-D-Glucans level in patients with Juvenile Idiopathic Arthritis | one year
  (1-3)-ß-D-Glucan (BDG), a component of most fungal cell walls, possess immunomodulatory activities. Latest studies demonstrate that it acts as a trigger for autoimmune arthritis in adult. BDG assays (Fungitell®) will be performed on serum of each JIA patients.

SECONDARY OUTCOMES:
Correlation of (1,3)-Beta-D-Glucans level in patients with Juvenile Idiopathic Arthritis score (JADAS) | one year
  The JADAS includes the following four measures: physician's global assessment of disease activity, measured on a 0-10 visual analog scale (VAS) where 0 = no activity and 10 = maximum activity; parent global assessment of well-being, measured on a 0-10 VAS where 0 = very well and 10 = very poor; the erythrocyte sedimentation rate (ESR), normalized to a 0 to 10 scale; and a count of joints with active disease.

CONTACTS AND LOCATIONS:
Overall Officials: Djamal-Dine Djeddi, MD, Principal Investigator — CHU Amiens; Taieb Chouaki, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No